CLINICAL TRIAL: NCT07198776
Title: Unilateral Versus Bilateral Vertebroplasty in Local Anaesthesia: A Prospective Randomised Comparative Study With 6-Month Follow-Up
Brief Title: Unilateral Versus Bilateral Vertebroplasty in Local Anaesthesia
Acronym: UNI-BI PVP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Igor Movrin (Other)
Responsible Party: Sponsor-Investigator, Igor Movrin, Professor of Surgery, University Medical Center Maribor, University Maribor
Organization: University Maribor (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: National Medical Ethics Commit
Record Dates: First submitted 2025-09-15; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Osteoporotic Vertebral Compression Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral Vertebroplasty (Experimental): Patients undergo percutaneous unilateral vertebroplasty with polymethylmethacrylate (PMMA) cement under local anaesthesia.
  Interventions: Procedure: Percutaneous Vertebroplasty
- Bilateral Vertebroplasty (Active Comparator): Patients undergo percutaneous bilateral vertebroplasty with polymethylmethacrylate (PMMA) cement under local anaesthesia.
  Interventions: Procedure: Percutaneous Vertebroplasty

INTERVENTIONS:
Procedure: Percutaneous Vertebroplasty — Injection of PMMA cement into fractured vertebra under fluoroscopic guidance.

SUMMARY:
Osteoporotic vertebral compression fractures are a common cause of severe back pain and disability in elderly patients. Percutaneous vertebroplasty (PVP) with polymethylmethacrylate (PMMA) cement is widely used to relieve pain and stabilize the fractured vertebra. However, there is ongoing debate whether unilateral or bilateral vertebroplasty provides better clinical and radiological outcomes. This prospective randomized controlled trial was conducted at the University Medical Center Maribor to compare unilateral versus bilateral PVP performed under local anaesthesia. A total of 196 patients with acute osteoporotic vertebral compression fractures were enrolled and randomly assigned to one of the two groups. The primary outcome measure was pain reduction assessed by Visual Analogue Scale (VAS). Secondary outcomes included functional improvement measured by the Oswestry Disability Index (ODI), procedure duration, fluoroscopy time, injected cement volume, radiological changes (vertebral height, kyphotic angle), and perioperative complications. The results are expected to provide evidence to guide optimal surgical management of osteoporotic vertebral fractures.

ELIGIBILITY:
* Age ≥65 years
* Single-level painful osteoporotic vertebral compression fracture (OVCF) confirmed radiologically
* Acute fracture (<6 weeks)
* Failure of conservative therapy
* Ability to provide written informed consentlusion Criteria:

Exclusion Criteria:

* Active infection
* Coagulopathy
* Burst fracture with retropulsion
* Neurological deficit
* Malignancy-related fracture

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 196 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity (VAS score) | From baseline (preoperative) to 6 months post-procedure
  Pain intensity measured on a Visual Analogue Scale (0-10; higher scores = worse pain).
Oswestry Disability Index (ODI) | From baseline to 6 months post-procedure
  Oswestry Disability Index score, range 0-100%, higher scores = greater disability.

SECONDARY OUTCOMES:
Operative time | During procedure
  Duration of vertebroplasty procedure measured in minutes.
Fluoroscopy time | During procedure
  Duration of fluoroscopic exposure during vertebroplasty, measured in seconds.
Injected cement volume | During procedure
  Total volume of polymethylmethacrylate (PMMA) cement injected into the fractured vertebra, measured in milliliters.
Vertebral height restoration | From baseline (preoperative) to hospital discharge (postoperative day 1)
  Percentage restoration of anterior vertebral body height on lateral radiographs.
Kyphotic angle correction | From baseline (preoperative) to hospital discharge (postoperative day 1)
  Change in local kyphotic angle (°) on lateral radiographs.
Complications | Intraoperative and 6 months post-procedure
  Incidence of perioperative and follow-up complications, including cement leakage, adjacent fractures, infection, or neurological events.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Maribor, Department of Traumatology, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: No